CLINICAL TRIAL: NCT00757263
Title: A Population Based Study of Genetic Predisposition and Gene-Environment Interactions in Ovarian Cancer in East Anglia, Oxford, Trent and West Midlands
Brief Title: Study of Genes and the Environment in Patients With Ovarian Cancer in the East Anglia, Oxford, Trent, or West Midlands Regions of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598881; MREC-SEARCH-OVARIAN; MREC-07/MRE05/17
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer; ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility for cancer and interactions between genes and the environment in patients with ovarian cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain epidemiological information and biological material on a population-based series of ovarian cases.
* To define the proportion of ovarian cancer incidence attributable to mutations in known predisposing genes (e.g., BRCA1 and BRCA2).
* To determine the risk associated with predisposing mutations by examining the cancer risks in relatives of patients who are shown to be carriers.
* To examine the effect of nongenetic risk factors in mutation carriers.
* To determine the pathological and clinical characteristics of ovarian cancers occurring in BRCA1/2 mutation carriers as compared with that in noncarriers.
* To establish whether mutations at other loci may predispose to ovarian cancer by comparing the frequency of alterations in ovarian cancer patients with that in cancer-free controls identified through the European Prospective Investigation of Cancer (EPIC) study.

OUTLINE: This is a multicenter study.

Patients complete an epidemiological questionnaire. The questionnaire will request identifying information on the patient's first-degree relatives.

Blood samples are collected from patients. DNA is extracted from these blood samples and from samples collected from cancer-free control participants in MREC-SEARCH-CONTROL as well as from additional controls through the European Prospective Investigation of Cancer (EPIC) study (a population based study of diet and health based in Norfolk, East Anglia). DNA samples are analyzed for polymorphisms of low penetrance cancer susceptibility genes.

In addition to the ovarian cancer patients recruited for this study, patients with breast, endometrial, prostate, colorectal, bladder, kidney, pancreatic, brain and esophageal cancer, malignant melanoma, and lymphoma cancer are recruited in the following related clinical trials: MREC-SEARCH-BREAST, MREC-SEARCH-ENDOMETRIAL, MREC-SEARCH-PROSTATE, MREC-SEARCH-COLORECTAL, and MREC-SEARCH-CANCER.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ovarian cancer within the past 5 years
* Identified through the East Anglia, Stoke and West Midlands Cancer Registries serving any of the following geographic regions of the United Kingdom:

  * East Anglia
  * Oxford
  * Trent
  * West Midlands

PATIENT CHARACTERISTICS:

* Identified by the patient's general practitioner as fit to contact for this study
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of epidemiological information and biological material
Proportion of ovarian cancer incidence attributable to mutations in known predisposing genes (e.g., BRCA1 and BRCA2)
Risk associated with predisposing mutations
Effect of nongenetic risk factors in mutation carriers
Pathological and clinical characteristics of ovarian cancers occurring in BRCA1/2 mutation carriers as compared with that in noncarriers
Exploration of mutations at other loci that may predispose to ovarian cancer

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom